CLINICAL TRIAL: NCT05799222
Title: Feasibility Study of an Intensive Nutrition Therapy Program for Improvement of Obesity and Diabetes in a Low-income Population
Brief Title: Medically Intensive Nutrition Therapy Program for Obesity and Diabetes in a Low-income Population
Acronym: MINT
Status: Recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Chika V. Anekwe, MD, MPH, Instructor in Medicine, Massachusetts General Hospital
Other Study IDs: 2022P001451
Record Dates: First submitted 2023-03-03; First posted 2023-04-05 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Overweight; PreDiabetes; Diabetes Type 2; Obesity
MeSH Terms: conditions — Overweight; Prediabetic State; Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Participants may choose to take part in an optional collection of stored blood.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults with overweight/obesity and pre-diabetes/diabetes and low income: Adults with overweight or obesity and pre-diabetes or type 2 diabetes who earn a low income.
  Interventions: Dietary Supplement: Bariatrix Meal Replacement Products

INTERVENTIONS:
Dietary Supplement: Bariatrix Meal Replacement Products — Meal replacement products offered through the Massachusetts General Hospital Weight Center.

SUMMARY:
This study is being done to better understand whether meal replacements can be an effective tool for weight loss and treatment of elevated blood sugars in people with obesity/overweight and diabetes/pre-diabetes who have a low income.

DETAILED DESCRIPTION:
The Medically Intensive Nutritional Therapy (MINT) program at Massachusetts General Hospital (MGH) Weight Center is a low-calorie nutrition plan that may offer a solution for those who have difficulty implementing a low-calorie dietary plan on their own. This study examines the effects of MINT on weight loss and blood sugar control specifically in a low-income population and explores potential reasons for discontinuing the program.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* Body mass index (BMI) greater than or equal to 27 kg/m^2
* HgA1C greater than or equal to 5.7 percent or fasting glucose greater than or equal to 100mg/dL within the previous 6 months
* Low-income as defined by having a family income at or below 400 percent of the federal poverty level guidelines for 2022

Exclusion Criteria:

* Current use of antihyperglycemic agents (other than metformin) or approved anti- obesity medications or plans to start such regimens over the 3 months post-study enrollment
* HbA1c greater than or equal to 10 percent
* Plans to pursue bariatric surgery over the 6 months post-study enrollment
* Weight loss of greater than 5 kg within the previous 3 months
* Current active eating disorder, with the exception of binge eating disorder
* Severe active psychiatric disease or significant cognitive impairment deemed by investigator likely to impede adherence to piloted intervention
* Active illicit substance abuse
* Pregnant, breastfeeding, or considering pregnancy within the next 6 months
* Current participation in another clinical research trial deemed by investigator to conflict with current study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with overweight or obesity and pre-diabetes or diabetes and low income
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-03-28 (Actual); Primary Completion 2026-11-08 (Estimated); Study Completion 2026-11-10 (Estimated)

PRIMARY OUTCOMES:
Body weight reduction | 3 months
  Reduction in body weight by greater than or equal to 5 percent
Hemoglobin A1c reduction | 3 months
  Reduction of Hemoglobin A1c by greater than or equal to 0.5 percent

SECONDARY OUTCOMES:
Program adherence | 3 months
  Adherence with the program, and potential reasons for non-adherence as assessed with bi-weekly questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Chika V Anekwe, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
There is no IPD plan.